CLINICAL TRIAL: NCT00457548
Title: Study of Effectiveness of BI Given to Injured MVC ED Patients Who Use Alcohol Harmfully and Hazardously
Brief Title: Phone Intervention for Alcohol (ETOH) Use in Emergency Department Motor Vehicle Crash (ED MVC) Patients
Acronym: DIAL
Status: Available | Type: Expanded Access
Sponsor: Rhode Island Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Michale Mello MD MPH, Rhode Island Hospital
Other Study IDs: R49/CCR123228-03
Record Dates: First submitted 2007-04-05; First posted 2007-04-06 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2009-02

CONDITIONS: Alcoholic Intoxication; Wounds and Injuries
Keywords: Alcohol use; Brief Interventions; Injuries; Emergency Department Patients; Harmful and hazardous alcohol use among ED injured patients
MeSH Terms: conditions — Alcoholic Intoxication; Wounds and Injuries; Alcohol Drinking

INTERVENTIONS:
Behavioral: Brief Telephone Counseling for risky aclohol use — Two brief sessions (30-40 minutes) of brief counseling using a motivational interviewing approach. The counseling session are delivered by telephone and focus on the alcohol use of inuured ED patients who randomize into the treatment arm of the study. Patient who randomize into the controla rm of the study receive standard emergency department care only plus study assessments.

SUMMARY:
The purpose of this study is to determine if a brief counseling intervention, delivered by telephone, is more effective than standard ED care, to reduce future alcohol related injuries and alcohol related negative consequences, among patients treated in the ED for injuries from an MVC and other injury mechanisms.

DETAILED DESCRIPTION:
Alcohol related motor vehicle crashes (MVC) continue to be a substantial public health problem. Brief interventions for alcohol (BI) for injured ED patients have been demonstrated to be effective, and perhaps more so for MVC patients.

Telephone interventions have been utilized in varying ways in health care. We compared the delivery of two brief interventions by telephone against an assessment only condition. Participants who received the BI and the assessment only condition were contacted 3 and 12 months after recruitment. Data about alcohol use, injuries and high risk behaviors, including drinking and driving behaviors were collected at the 3 and 12 month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Emergency department patient
* Subacute injury
* Motor vehicle crash or other injury
* Alcohol use at harmful and hazardous levels

Exclusion Criteria:

* Younger than 18 years old
* Does not meet alcohol use criteria
* Non-English speaker
* In police custody
* Suicidal
* Psychiatric diagnosis
* No locator
* Injury occurred > 72 hours prior to ED visit

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Mello MJ, Longabaugh R, Baird J, Nirenberg T, Woolard R. DIAL: a telephone brief intervention for high-risk alcohol use with injured emergency department patients. Ann Emerg Med. 2008 Jun;51(6):755-64. doi: 10.1016/j.annemergmed.2007.11.034. Epub 2008 Apr 23. PMID 18436341